CLINICAL TRIAL: NCT03317340
Title: Environmental Factors to Increase Patient Comfort During Urodynamics Testing
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Aqsa A. Khan, Principle Investigator, Mayo Clinic
Other Study IDs: 17-003351
Record Dates: First submitted 2017-10-03; First posted 2017-10-23 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Lower Urinary Tract Symptoms; Urologic Diseases
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient Undergoing Urodynamics
  Interventions: Other: Background Sounds

INTERVENTIONS:
Other: Background Sounds — Background music or sound of running water

SUMMARY:
Urodynamics is a comprehensive study of the lower urinary tract. Although the information obtained from urodynamics answers several questions and assists in guiding therapies for patients, the testing environments is unnatural and may be distressing for patients. This may impact the results of the study, as it is not uncommon for patients to be unable to void for the test due to their distress. Often to alleviate the distress, music or soothing noises are used in the background. The study aims to identify simple environmental factors which may improve patient experience with urodynamic testing. The population will include patients with existing appointments for urodynamics testing at the Mayo Urology Clinic. The investigators plan to assess patient satisfaction and comfort during this assessment using a visual analog scale questionnaire. The environmental variables will include music of the patients' preference, the sound of running water, or no background noise at all. By asking patients to complete a questionnaire, The investigators will be able to assess ways to improve patient comfort in a commonly used urologic assessment.

ELIGIBILITY:
Inclusion Criteria:

* All adults undergoing urodynamics
* Must be able to understand and complete questionnaire

Exclusion Criteria:

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing urodynamics
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Comfort level with test based off post-urodynamic survey | 6 months
  visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Aqsa A Khan, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials